CLINICAL TRIAL: NCT00613613
Title: The Impact of Genetic Determinants of Fenofibrate's Pharmacogenetics on Lipid Response
Brief Title: Fenofibrate and Pharmacogenetic Impact in Dyslipidemia
Acronym: FPI
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: 0708M15441; AHA Grant #0755839Z (Other: University of Minnesota)
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: High drug metabolism genotype All receive fenofibrate
  Interventions: Drug: fenofibrate
- 2: Low drug metabolism genotype All receive fenofibrate
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate — Fenofibrate 145mg tablets once daily for 4 weeks
  Other Names: TriCor® 145mg tablets
  Groups: 1
Drug: fenofibrate — Fenofibrate 145mg tablets once daily for 4 weeks
  Other Names: TriCor® 145mg tablets
  Groups: 2

SUMMARY:
The purpose of the study is to learn whether genetics plays a role in predicting response to a commonly used and FDA (Food and Drug Administration) approved medication for lowering triglycerides and cholesterol. The hypothesis: The pharmacogenetics of genes which affect drug metabolism (how the body handles the drug) and drug targets (how the drug acts on the body) influences how a person responds to the lipid lowering medication-fenofibrate.

DETAILED DESCRIPTION:
The investigators seek to screen over 200 subjects for select candidate genes to serve as a source of subjects which may participate in a genotype guided investigation as to the predictability of response based on genotype. Response endpoints relate to lipid parameters and other variables of interest to cardiovascular endpoints. Subjects with genotypes of interest would then be enrolled into a short term clinical trial evaluating their response to fenofibrate based on their genetic profile ascertained from the screening phase.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year old
* Be willing to participate in the study and attend the scheduled clinic exams
* Consent to taking lipid lowering therapy for 4 weeks and if necessary discontinue lipid lowering agents for a period of 8 weeks

Exclusion Criteria:

* <18 years of age
* History of liver, kidney, pancreas, pancreatitis, gall bladder disease or malabsorption (Crohn's disease etc.)
* Use of insulin or currently taking warfarin
* Pregnant women or women of childbearing potential not using an acceptable form of contraception
* History of an allergy or hypersensitivity to fenofibrate
* Investigational drug use within 30 days of the study
* A disease that, in the opinion, of the PI, would put the subject at risk during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with dyslipidemia
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- serum concentration of fenofibric acid AUC (0-24hrs) for high vs low metabolizers | 24 hours
  We measured area under the curve (AUC) in mcg*hr/mL (from time 0 to 24 hrs) at steady state for those of two specific genotypes for our UGT2B7 SNP following steady-state dosing of fenofibrate.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Straka, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States